CLINICAL TRIAL: NCT01588314
Title: Placebo Controlled Trial Evaluating Gabapentin for the Treatment of Small Fiber Neuropathic Pain in Patients With Fabry Disease
Brief Title: Safety and Efficacy of Gabapentin for Neuropathic Pain in Fabry Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients were enrolled. No data & no study results to report.
Sponsor: University of Minnesota (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1112M07943
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Fabry Disease; Neuropathic Pain
Keywords: Fabry disease; neuropathic pain; gabapentin
MeSH Terms: conditions — Fabry Disease; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gabapentin (Active Comparator)
  Interventions: Drug: Gabapentin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Gabapentin — gabapentin 100 mg capsules
  Other Names: Neurontin
  Arms: gabapentin
Drug: placebo — compounded placebo capsules
  Arms: placebo

SUMMARY:
The purpose of this study is to determine efficacy of gabapentin vs. placebo at controlling peripheral neuropathic pain in patients with Fabry disease, and reducing their use of opioid analgesics. The investigators are conducting a randomized, double-blind, placebo controlled, single center, cross-over study. The primary endpoint is percent reduction in patients' use of hydrocodone-acetaminophen.

DETAILED DESCRIPTION:
Fabry disease is an X-linked lysosomal storage disorder which results from reduced activity of the enzyme α-galactosidase A. This reduced enzyme activity results in accumulation of globotriaosylceramide (GL-3), which causes disturbances in multiple organ systems. Patients often complain of acroparesthesia, caused by small-fiber neuropathy. Limited information is available regarding effective treatments for small-fiber neuropathic pain in Fabry disease, and no standard-of-care has yet been established. Opioid analgesics are often used because of their pharmacokinetic properties. While effective, the use of opioids has complications such as constipation, physical dependence and addiction. The purpose of this study is to determine efficacy of gabapentin vs. placebo at controlling peripheral neuropathic pain and reducing the use of opioid analgesics. The investigators are conducting a randomized, double-blind, placebo controlled, single center, cross-over study. The primary endpoint is percent reduction in hydrocodone-acetaminophen use.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Fabry Disease
* age ≥ 18 years of age at study enrollment
* current neuropathic pain at any severity level

Exclusion Criteria:

* known sensitivity or allergy to study drug
* history of illicit drug use
* pregnancy
* suicidal thoughts at study enrollment as assess by the C-SSRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
average reduction in hydrocodone-acetaminophen use | assessed at the end of the study

SECONDARY OUTCOMES:
Number and type of adverse events | assessed at the end of the study
Pain levels | assessed at the end of the study
Define therapeutic level for gabapentin | assessed at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine R. Jarnes, PharmD, Principal Investigator — University of Minnesota, Fairview
Locations (1):
- University of Minnesota, Fariview, Minneapolis, Minnesota, United States